CLINICAL TRIAL: NCT04998344
Title: An Effectiveness Trial (Phase IV) to Evaluate Protection of Children and Pregnant Women by Influenza Vaccine in Rural Bangladesh
Brief Title: An Effectiveness Trial to Evaluate Protection of Children and Pregnant Women by Influenza Vaccine in Rural Bangladesh
Acronym: FluEffect
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Rebecca Cox, Professor Rebecca Cox, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR-19103
Record Dates: First submitted 2021-04-26; First posted 2021-08-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Influenza Viral Infections
Keywords: influenza; vaccine; safety; immunogenicity; effectiveness
MeSH Terms: conditions — Influenza, Human | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inactivated influenza vaccine group (Experimental): Vaccines will be administered as a single dose regimen for the pregnant women and two doses for children at 28-day interval as recommended by the vaccine manufacturers.
  Interventions: Biological: Inactivated influenza vaccine
- Inactivated polio vaccine group (Active Comparator): Vaccines will be administered as a single dose regimen for the pregnant women and two doses for children at 28-day interval as recommended by the vaccine manufacturers.
  Interventions: Biological: Inactivated polio vaccine

INTERVENTIONS:
Biological: Inactivated influenza vaccine — Vaccines will be administered as a single dose regimen for the pregnant women and two doses for children at 28-day interval as recommended by the vaccine manufacturers.
  Arms: Inactivated influenza vaccine group
Biological: Inactivated polio vaccine — Vaccines will be administered as a single dose regimen for the pregnant women and two doses for children at 28-day interval as recommended by the vaccine manufacturers.
  Arms: Inactivated polio vaccine group

SUMMARY:
Annually influenza is a leading cause of severe disease and mortality particularly in young children <5 years old and pregnant women in the low and middle-income countries (LMICs) and both groups are prioritised for vaccination by the World Health Organisation (WHO). In Bangladesh, influenza is responsible for 10% of all childhood pneumonias and 9% of all death. Maternal influenza is associated with an increased risk of hospitalisation and foetal malformation. Influenza is a vaccine preventable disease, however, in most LMICs influenza vaccination is not part of the vaccination programme. This study will evaluate the effectiveness of inactivated influenza vaccine against influenza illness among pregnant women and children in Bangladesh. Influenza vaccine has not yet been studied as combined immunization strategy in a cluster randomized trial. This study is a community-based randomised trial in both pregnant women and young children to assess the impact of inactivated influenza vaccine in preventing influenza in the community as well as population level impact by both direct and indirect effect of vaccination.

DETAILED DESCRIPTION:
This clinical trial will be conducted in rural Matlab, Bangladesh, covered by a Maternal, Child Health and Family Planning intervention program (named MCH-FP area). Twenty villages in the Maternal, Child Health and Family Planning intervention program area will be randomized at a 1:1 ratio to receive either inactivated influenza vaccine (IIV) or the control inactivated polio vaccine (IPV). Recruitment, randomization and vaccination of healthy pregnant women at 28 to 34 weeks of gestation period and children 6 to 59 months old at the time of enrolment will be carried out from fixed site clinics working in the MCH-FP area. Vaccines will be administered as a single dose regimen for the pregnant women and two doses for children at 28-days interval as recommended by the vaccine manufacturers. All pregnant women in the third trimester of pregnancy (n~300), and children 6 to 59 months old in 20 villages in the MCH-FP area of Matlab will be eligible for vaccination (n~3500) for the study. In addition, all residents of study villages will be included in the influenza surveillance.

All vaccinated pregnant women and parents of vaccinated children 6 to 59 months old will be asked to inform the study team by phone of any respiratory illnesses or to visit the Matlab hospital. Also, all residents of the study villages will be asked to visit the Matlab hospital/fixed site clinic for any respiratory illness. Participants will receive regular SMS messages to remind them to report cases of influenza like illness (ILI). At the hospital, the medical officer will examine the sick patient and decide if the criteria of the ILI case definition are met. ILI is defined as an acute respiratory infection with: measured fever of ≥ 38 C° and cough; with onset within the last 10 days for adults; and in case of children as measured axillary temperature ≥ 38.0°C with onset within the last 10 days and at least one of the following symptoms: cough, sore throat, nasal congestion, rhinorrhea, earache or ear discharge. In medically confirmed ILI cases, the trial will collect nasopharyngeal and throat swabs for confirmation of the aetiology of the infection, as well as collect serum samples from vaccinated participants Passive surveillance will continue for 18 months following completion of vaccination.

Outcome measures/variables:

1. Incidence, prevalence, seasonality and clinical descriptions of :

   1. Influenza infection including clinical pneumonia in child (fever, cough and respiratory difficulties)
   2. Influenza infection including clinical pneumonia in mother (fever, cough and respiratory difficulties)
2. HAI antibody titres to calculate the rate of reduction of risk of influenza infection or disease in influenza vaccination pregnant women and children as well as reduction of flu infection in population of intervention and control villages
3. Evaluation of simple sample collection methods in children to assess Influenza specific antibody responses in DBS and saliva sample
4. Clinical and demographic risk factors associated with illness
5. Comparisons of pregnancy outcomes and post-delivery illness/complication
6. Clinical and laboratory confirmation of influenza and other respiratory virus in sick individuals
7. Economic evaluation of influenza vaccination in pregnant women and children

ELIGIBILITY:
Inclusion Criteria for Pregnant women:

* Permanent Resident in selected villages in Matlab HDSS MCH-FP area
* Age 18 - 49 years old
* 28 to 34 weeks of gestation at the time of enrollment
* Willing to stay in the study village for the next 20 months

Exclusion Criteria for Pregnant Women:

* Refusal to provide consent for participation
* Unable to participate in the full length of the study period
* Known allergy to egg or any product of vaccine
* Sick (has documented fever and respiratory illness) at the time of enrollment
* Pregnancy with complications such as chronic pulmonary (including asthma), cardiovascular, renal, hepatic, hematologic (including sickle cell disease), or metabolic disorders (including diabetes mellitus and obesity) or neurologic and neurodevelopment conditions, cancer, immunosuppression, and, multiple pregnancy)
* Received any vaccine /immune component in last 2 weeks
* Participated in any research study in the last 3 months

Inclusion Criteria for Children:

* Permanent Resident in selected villages in Matlab HDSS MCH-FP area
* Age 6 to 59 months old
* Parents/guardians confirm their willingness to stay in the study village for the next 20 months

Exclusion Criteria for Children:

* Parents refuse to provide consent for participation
* Unable to participate in the full length of the study period
* Known allergy to egg or any product of vaccine
* Sick children (has documented fever and respiratory illness) at the time of enrolment
* Chronic illness such as chronic pulmonary (including asthma), cardiovascular, renal, hepatic, hematologic (including sickle cell disease), or metabolic disorders (including diabetes mellitus and obesity) or neurologic and neurodevelopment conditions, cancer, and immunosuppression
* Received any vaccine /immune component in last 4 weeks
* Participated in any research study in the last 3 months

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3800 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of influenza vaccination in reducing rates of acute respiratory infections due to laboratory-confirmed influenza in pregnant women at 28 to 34 weeks of gestation period and children 6 to 59 months old | through study completion, an average of 3 year
  The direct effectiveness of influenza vaccine in reducing rates of acute influenza infections in vaccinated patients attending a treatment facility will be assessed. The indirect effectiveness will be calculated by comparing the rates of influenza in the villages where influenza vaccine is introduced to the influenza rates in people from villages vaccinated with the control vaccine.

SECONDARY OUTCOMES:
Safety of influenza vaccine among pregnant women at 28 to 34 weeks of gestation period and children 6 to 59 months old in Bangladesh | through study completion, an average of 1.5 year
  The safety of the vaccine will be monitored through a field visit on Day 3 after each dose of vaccination and thereafter by telephone. All adverse events will be recorded, and any serious adverse events will be investigated. Adverse events after vaccination will be summarized and compared between the intervention and control groups.
Surveillance for influenza and other respiratory viruses | through study completion, an average of 3 year
  In medically confirmed ILI cases, nasopharyngeal and throat swabs will be collected for laboratory confirmation of the aetiology of the infection, Passive surveillance will continue for 18 months following completion of vaccination.
Vaccine immunogenicity in pregnant women and children | through study completion, an average of 3 year
  The hemagglutination inhibition assay will be used to assess the vaccine immunogenicity to the homologous vaccine strains and appropriate epidemic strains.
Indirect vaccine effectiveness of influenza vaccination of pregnant women and children | through study completion, an average of 3 year
  All residents of the 20 study villages will be included in the influenza surveillance. Influenza cases will be defined as laboratory confirmed rRT-PCR influenza A and/or B viruses during the influenza surveillance period. The total and indirect vaccine protection in the population will be assessed from medical records for birth outcomes, birth weights, ILI, hospitalization and death records in Matlab.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Cox, PhD, Principal Investigator — University of Bergen, Norway
Locations (2):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: icddr, b is an international health research organisation located in Dhaka, Bangladesh — https://www.icddrb.org/
- See also: The Influenza Centre is a collaboration between the University of Bergen, The Haukeland University Hospital and the Department of Health. — http://www.influensasenteret.no/